CLINICAL TRIAL: NCT05690464
Title: Trial of Magnesium Supplementation and Blood Pressure Reduction Among Adults With Elevated Systolic Blood Pressure
Brief Title: Effect of Magnesium Supplementation on Elevated Systolic Blood Pressure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Pure Encapsulations (Industry)
Responsible Party: Principal Investigator, Howard D. Sesso, ScD, MPH, Associate Epidemiologist, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022P002101
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Blood Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- magnesium (Active Comparator): magnesium glycinate supplement, 480 mg/day
  Interventions: Dietary Supplement: magnesium glycinate supplement
- placebo (Placebo Comparator): placebo supplement
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: magnesium glycinate supplement — magnesium glycinate (480 mg/day)
  Arms: magnesium
Dietary Supplement: placebo — placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to assess whether 480 mg/day magnesium glycinate supplementation for 12 weeks lowers blood pressure.

DETAILED DESCRIPTION:
This clinical trial will test whether a magnesium glycinate supplement (480 mg/day) taken for 12 weeks lowers blood pressure in 120 adults aged 30-74 who have a systolic blood pressure of 130-154 mmHg.

Eligibility to participate in the trial will be determined by a 2-stage screening process. Interested participants will complete a pre-screening form online. If eligibility criteria are met, the potential participants will be scheduled for an in-person screening clinic visit. At the visit, eligible participants will be reminded about the study details and potential risks and will be given the opportunity to sign the Informed Consent. Consented participants will be assigned by chance (like a coin toss) to daily magnesium or to placebo. Participants will take 4 study capsules per day (2 capsules in the morning and 2 capsules in the evening) for 12 weeks.

Assessments at the screening visit include seated blood pressure; pulse; weight, height, waist and hip circumference measurements; fasting blood and urine collection; and health and diet questionnaires. Participants will return for a clinic visit at 12 weeks to assess these measures.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of systolic blood pressure 125-159 mmHg
* Measured seated systolic blood pressure 130-159 mmHg at screening visit
* Body mass index less than 40 kg/m2
* Total magnesium intake from supplements of no more than 100 mg/day
* Willing to maintain current diet and supplement use patterns during the 12-week intervention period

Exclusion Criteria:

* Measured seated diastolic blood pressure 100 mmHg or greater at screening visit
* Antacid or laxative use 4 times/week or more within the past 3 months
* History of cardiovascular disease (myocardial infarction, stroke, revascularization [coronary artery bypass graft or percutaneous transluminal coronary angioplasty], or angina pectoris)
* History of invasive cancer diagnosed within the last 5 years (non-melanoma skin cancer permitted)
* History of type 1 or 2 diabetes
* History of renal disease
* History of kidney failure
* History of dialysis
* History of pancreatitis
* History of inflammatory bowel disease
* History of hypermagnesemia
* Women who are pregnant, nursing, or intend to become pregnant during the period of treatment
* Plan to relocate out of Boston area within the next year
* Unwillingness and/or inability to swallow 4 pills per day
* Inability to provide written informed consent

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in seated systolic blood pressure from baseline to 12 weeks | Baseline and 12 week
Change in seated diastolic blood pressure from baseline to 12 weeks | Baseline and 12 week

SECONDARY OUTCOMES:
Change in serum magnesium levels from baseline to 12 weeks | Baseline and 12 week
Change in RBC magnesium levels from baseline to 12 weeks | Baseline and 12 week
Whether the effect of magnesium on seated blood pressure is modified by baseline serum and/or RBC magnesium | Baseline and 12 week

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No